CLINICAL TRIAL: NCT02304978
Title: Prognostic Value of Tissue Factor (TF) in Blood t in Colorectal Cancer in Adults
Acronym: TF
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-09/0908; 2009-A00264-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-06-24; First posted 2014-12-02 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Tissular factor; TF
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CRC (Experimental): patient with a colorectal cancer
  Interventions: Biological: Group CRC
- Group control (Experimental): Control - volunteers
  Interventions: Biological: Group control

INTERVENTIONS:
Biological: Group CRC — blood samples
  Arms: Group CRC
Biological: Group control — Blood samples
  Arms: Group control

SUMMARY:
Severity of colorectal cancer (CRC) is evaluated by its local staging, locoregional and general ( presence of metastases , usually liver ). This is the most common cancer in France and, despite surgical treatment of the primary tumor, it is still subject to a high mortality rate due to metastatic evolution, mainly hepatic .

There is currently no specific marker for predicting cancer, the same hardly changed , which would modulate the aggressive therapeutic strategy . antigen (CEA) is used in the monitoring of JRC made.Tissue factor (TF) is the VII tissue factor receptor. it initiates the coagulation cascade. it was noted as a true cell marker tumorale1 aggressiveness. Corroborating evidence that the way the TF plays an important role in the invasive and metastatic potential of CRC. First, various human cancer cell lines express the FT colic. Furthermore, there is a relationship between the importance of monocyte TF expression and the evolutionary potential of human CRC.

The investigators hypothesize that these interest intra-platelet and plasma markers are a reflection of tumor angiogenic potential. And the investigators will verify the superiority of their preoperative levels in the CRC group compared with the control group, normalization of postoperative after surgical resection rates and their possible re-ascent in case of tumor recurrence in the CRC group.

The levy to one month in controls allow us to verify the absence of secondary modification to laparotomy, the colectomy and general anesthesia.

The investigators assume that the rate of soluble TF in peripheral blood of the holders of CRC patients may be a marker of invasion and aggression (i.e. prognosis).

DETAILED DESCRIPTION:
The study is to measure the TF in the blood, as well as ACE, C reactive protein and E-selectin. The TF will also be measured in the tissue removed during surgery.

ELIGIBILITY:
Inclusion Criteria:

All patients, adults, holders of CRC with or without MH in whom surgical resection HEALING is planned .

For witnesses:

- Patients without CCR (preoperative colonoscopy). This control population will verify normal values regulators of angiogenesis recently defined and specificity of these vis-à-vis markers CCR-

Exclusion Criteria:

all situations where the plasma levels of FT antigen are high, in particular:

* Patients with unstable angina or myocardial infarction in the acute phase (not older than two months)
* Severe sepsis (hospitalization)
* Cirrhosis stage Child C
* Chronic renal failure requiring renal replacement extra
* Patients with microvascular complications of diabetes
* Vasculitis
* Pregnancy and lactation patient on oral contraceptives, or having hormone replacement therapy for menopause

  * Patients with extrahepatic metastases
  * Patients underwent emergency surgery
  * Persons not able to consent

For witnesses:

History of cancer, inflammatory disease, diabetes, regular intake of anti inflammatory drugs.

If during colonoscopy, colorectal cancer was detected, the control patients were excluded from the study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-06-22 (Actual); Primary Completion 2015-05-26 (Actual); Study Completion 2015-05-26 (Actual)

PRIMARY OUTCOMES:
TNM primary colorectal tumor stage | Before surgery
  soluble blood TNM value will be determined before surgery, and compared between groups.

SECONDARY OUTCOMES:
TF (blood levels of soluble TF) | 1 , 6 , 12, 18 and 24 months .5 years
  Comparing the pre - operative and post -operative blood levels of soluble TF and TF intratumoral
TF intratumoral (blood levels of TF intratumoral) | 1 , 6 , 12, 18 and 24 months .5 years
  Comparing the pre - operative and post -operative blood levels of soluble TF and TF intratumoral
E- selectin and CRP | 1 , 6 , 12, 18 and 24 months. 5 years
  Comparison - soluble TF with blood levels of other circulating proteins: E- selectin and CRP at different times of follow-up.
ACE | 1 , 6 , 12, 18 and 24 months .5 years
  Evaluation of the prognostic value of blood levels of soluble TF and that of ACE blood on the incidence of Metastases Hepatic in patients undergoing CRC and / or hepatic
Interaction plate / tumor cell | 1 , 6 , 12, 18 and 24 months .5 years
  Quantifying the interaction plate / tumor cell by measuring intraplatelet regulatory proteins and angiogenesis markers of platelet activation and plasma compare the

CONTACTS AND LOCATIONS:
Overall Officials: ZERBIB Philippe, Prof, Study Director — CHRU of LILLE
Locations (1):
- Service de Chirurgie Digestive et de transplantation Hôpital Claude HURIEZ, Lille, France

IPD SHARING:
Plan to Share IPD: No